CLINICAL TRIAL: NCT02211768
Title: Transformation of Plexiform Neurofibromas to Malignant Peripheral Nerve Sheath Tumors in Neurofibromatosis Type 1: Clinical, Histopathologic, and Genomic Analysis
Brief Title: Transformation of Plexiform Neurofibromas to Malignant Peripheral Nerve Sheath Tumors in Neurofibromatosis Type 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 140163; 14-C-0163
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-07-23

CONDITIONS: Neurofibromatosis; MPNST
Keywords: Genetic Analysis; Biopsy; FDG-PET; FLT-PET
MeSH Terms: conditions — Neurofibromatoses; Neurofibrosarcoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/FDG and FLT PET scans (Experimental): Subjects will undergo FDG-PET and FLT-PET scans at least one day apart
  Interventions: Procedure: MRI, FDG-PET/CT scans; Drug: [18F]-FLT-PET/CT scans
- 2/FDG-PET scan (Other): Subjects will undergo FDG-PET scan
  Interventions: Procedure: MRI, FDG-PET/CT scans

INTERVENTIONS:
Procedure: MRI, FDG-PET/CT scans — Standard of care to be obtained as part of the study
Drug: [18F]-FLT-PET/CT scans — FLT PET to be performed as a research imaging study as it is not considered standard imaging in NF1
  Arms: 1/FDG and FLT PET scans

SUMMARY:
Background:<TAB>

- Many people with neurofibromatosis type 1 (NF1) get tumors of the nervous system. Finding malignant tumors early is important for removing them. Researchers want to find ways of doing this with scans and genetic testing.

Objectives:

- To learn more about neurofibromatosis type 1.

Eligibility:

- People age 10 and older with NF1 who have a benign tumor or have had a malignant one.

Design:

* Participants will be screened in another study with medical history, physical exam, and urine and blood tests. They will have a magnetic resonance imaging (MRI) scan.
* MRI: Participants will lie on a table that slides into a metal cylinder. They will be in the scanner for 60 90 minutes, lying still for 15 minutes at a time. Participants will get earplugs for the loud sounds. They will get a contrast agent (dye) through a thin plastic tube (catheter) inserted in an arm vein.
* As part of their regular care, participants will have:
* FDG-PET/CT scan. They will get radioactive glucose (sugar) through a catheter in an arm vein.
* [18F]-FLT-PET/CT scan. This is like the FDG scan but with a different radioactive chemical.
* Biopsy. A piece of tumor tissue is removed with a needle. A piece of tissue from a previous biopsy may also be studied.
* Participants may have genetic testing. Blood will be taken. It will be tested along with biopsy samples. Researchers will explain the risks and procedures. They may notify participants if testing shows health problems.
* After this study, participants will continue their regular cancer care.

DETAILED DESCRIPTION:
Background:

* NF1 is an autosomal dominant genetic disorder characterized by distinct features including the development of benign plexiform neurofibromas (PN) and malignant peripheral nerve sheath tumors (MPNST) tumors of the nervous system.
* Development of MPNST typically results from malignant transformation in a preexisting PN. Associated symptoms may overlap and be difficult to distinguish from growth of a benign PN. Currently surgery is the only standard treatment for PN and MPNST.
* The 5-year overall survival rate for NF1 patients with a MPNST is poor; therefore, early detection of malignant transformation of a PN is an important goal.
* Fluoro-deoxy-glucose (FDG) positron emission tomography (PET) in NF1 has utility in detecting malignant transformation. However, concerning lesions can have high FDG uptake and be benign on biopsy.
* Fluoro-thymidine (FLT) PET measures cell cycling and proliferation. Malignant lesions have higher proliferation rates than benign tumors; therefore, FLT-PET may be sensitive and specific in the early detection of malignant transformation and assess response.
* Genetic analysis is an important component in evaluating the transformation of PN to MPNST. Biallelic NF1 and tumor suppressor gene mutations (p53, INK4A, p27kip1), increased Ras activity and abnormal growth factor signaling have been described, but there is no known signature for MPNST.
* Massively parallel ( next generation ) sequencing technology permits whole-genome, whole-exome and transcriptome sequencing of multiple tumors including MPNST.

Objectives:

* Determine the feasibility of FLT PET in patients with NF1 and MPNST or lesions concerning for MPNST, or MPNST.
* Evaluate the ability of FLT PET to distinguish benign PN from malignant lesions, and to determine if FLT PET is more accurate than FDG PET in correctly classifying a tumor as benign or malignant.
* Evaluate the feasibility of whole-exome sequencing and other genetic/genomic methods, including detection of epigenetic and/or expression changes and RNA Seq of tumor (MPNST or lesion concerning for MPNST and adjacent benign PN) biopsies using interventional radiology sampling techniques in consenting individuals with NF1 participating in 10-C-0086.
* Perform detailed clinical analysis of individuals with NF1 and MPNST or lesions concerning for MPNST.
* Perform detailed pathologic analysis of biopsy specimens from tumor areas to determine if increased uptake of FDG or FLT predicts for malignant transformation.
* Identify somatic genetic variants that distinguish PN from MPNST and from germline sequence by whole-exome sequencing potentially identifying targets for treatment.

Eligibility:

* NF1 patients with lesions concerning for malignancy or with active MPNST.
* Willingness to enroll on NCI protocol 08-C-0079: Natural History Study and Longitudinal Assessment of Children, Adolescents, and Adults with Neurofibromatosis Type 1.

Design:

* Up to 15 patients will be enrolled on this pilot study.
* Patients will undergo the following evaluations:
* Detailed clinical evaluation of NF1 manifestations on NCI protocol #08-C-0079
* Imaging studies including:

  * MRI, FDG-PET/CT scans (as standard care) in all subjects; and
  * [(18)F]-FLT-PET/CT (research study) in subjects 10 years of age or older
* Genetic counseling (if participating in the germline blood sampling and biopsy analysis portion of the study)
* Tissue analysis:

  ---Patients 18 years of age or older with MPNST will participate in tissue analysis, if consenting and appropriately preserved archival tissue is available, or if patient agrees to optional research biopsy (if consented and safe). Patients with lesions concerning for malignancy will undergo clinically indicated biopsies of concerning lesions and of adjacent benign PN (if consented and safe) for detailed pathologic analysis and whole-exome sequencing (co-enrollment on 10-C-0086 Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies). Biopsies to be directed by PET fusion imaging in interventional radiology.
* Whole-exome sequencing of a germline blood sample (optional) if participating in the tissue analysis (co-enrollment on 10-C-0086 Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies).
* To better characterize lesions concerning for MPNST and predict those at higher risk for malignant transformation, we will correlate clinical and imaging findings, including radiographic evaluation with FDG-PET/CT, and [(18)F]-FLT-PET/CT, pathologic evaluation of tumor biopsies (if available), and analysis of whole exome sequencing of germline blood samples (if consented) and of tumor samples (when available).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age:
* No upper age limit for patient enrollment.

  * FLT PET: will only be performed in patients greater than or equal to 10 years old
  * Research biopsies in consenting patients with MPNST: will only be performed in patients greater than or equal to 18 years old

    2. Diagnosis:
* Patients who are diagnosed with NF1 using the NIH Consensus Conference criteria or have a confirmed NF1 mutation with analysis performed in a CLIA certified laboratory. NF1 mutation testing to confirm eligibility will not be performed on this protocol, but as part the POB separate screening study.
* For the clinical diagnosis of NF1 all study subjects must have at two or more diagnostic criteria for NF1 listed below (NIH Consensus Conference):

  1. Six or more caf(SqrRoot)(Copyright)-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects)
  2. Greater than or equal to 2 neurofibromas or 1 plexiform neurofibroma
  3. Freckling in the axilla or groin
  4. Optic glioma
  5. Two or more Lisch nodules
  6. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  7. A first-degree relative with NF1

  3. NFI tumor manifestations

Subjects must have:

1. Diagnosis of NF1 with a lesion concerning for MPNST

   -Criteria include pain, growth of a known plexiform neurofibroma, abnormality on functional imaging study (FDG-PET) or change in clinical exam.

   OR
2. Diagnosis of NF1 with a histologically confirmed MPNST.

4. Subjects must be eligible for and willing to participate and sign consent for NCI protocol 08-C-0079: Natural History Study and Longitudinal Assessment of Children, Adolescents, and Adults with Neurofibromatosis Type 1, for the clinical evaluation necessary for this study.

5. Prior and current therapy:

For NF1 related benign tumor manifestations there is no standard effective medical treatment, and surgery is the only standard treatment. Chemotherapy and radiation therapy are additional treatment options for malignant NF1 related tumors. For the purpose of this study subjects who have not previously received medical or surgical treatment, patients who have previously received medical or surgical treatment, and subjects who are currently receiving medical treatment and or radiation for a NF1 related manifestation will be eligible.

Patients must be recovered from acute toxicities of prior therapy in order to be able to safely undergo biopsies proposed on the trial. Prior and current treatment for NF1 related manifestations will be recorded on protocol 08-C-0079.

Prior radiation therapy and chemotherapy in patients with MPNST must not have been administered within 4 weeks prior to enrollment.

6. Performance Status:

ECOG less than or equal to 3. Subjects who are wheelchair bound because of paralysis will be considered ambulatory when they are up in their wheelchair. Subjects have to be able to travel to the NIH for evaluations.

7. Informed Consent:

All patients or their legal guardians (if the patients is<18 years old) must sign an IRB-approved document of informed consent to demonstrate their understanding of the investigational nature and the risks of this study before any protocol-related studies are performed. When appropriate, pediatric subjects will be included in all discussions.

8. Hematologic criteria (applicable only in patients undergoing biopsy)

* Platelet count has to be greater than or equal to 100,000/microL
* Patients should have INR<1.4 and PT less than or greater to 40 seconds (unless due to lupus anticoagulant). In patients not meeting these parameters, clearance by hematology will be required prior to undergoing biopsy.

EXCLUSION CRITERIA:

1. Allergy or relative contraindications to MRI contrast agents.
2. Patients who require sedation for imaging studies will be excluded from the FLT PET scan research test. They will undergo only the standard of care MRI and FDG PET scan.
3. Contraindication to MRI scanning, such as surgery that involves metal clips or wires or metal prostheses which might be expected to cause tissue damage or produce image artifacts.
4. Patients with severe chronic renal insufficiency (glomerular filtration rate < 30 mL/min/1.73 m(2)), hepatorenal syndrome or post-liver transplantation.
5. History of prior fluorothymidine allergy or intolerance.
6. Participants with severe claustrophobia not relieved by oral anxiolytic medication or patients weighing >136 kg (weight limit for scanner table)
7. Pregnant women are excluded from this study because of the effects of radioactive materials with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with radioactive materials, breastfeeding should be discontinued.
8. Requirement for medications, which interfere with platelet function, such as aspirin, which cannot be stopped within 1 week prior to the biopsy (applicable only to patients undergoing biopsy).

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of whole-exome sequencing and other genetic/genomic methods | 3 years
  Genomic profile of subject's tumors to catalogue mutations associated with the development of a PN and then a MPNST
Evaluate the ability of FLT PET to distinguish benign PN from malignant lesions, and to determine if FLT PET is more accurate than FDG PET in classifying a tumor as benign or malignant | 3 years
  Proportion of patients identified with benign or malignant tumor using FLT PET versus FDG PET
Determine the feasibility of FLT PET in patients with NF1 and lesions concerning for MPNST, or MPNST | 3 years
  Sensitivity of FLT PET in distinguishing benign from malignant lesions

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Benz MR, Czernin J, Dry SM, Tap WD, Allen-Auerbach MS, Elashoff D, Phelps ME, Weber WA, Eilber FC. Quantitative F18-fluorodeoxyglucose positron emission tomography accurately characterizes peripheral nerve sheath tumors as malignant or benign. Cancer. 2010 Jan 15;116(2):451-8. doi: 10.1002/cncr.24755. PMID 19924789
- [Background] Meany H, Dombi E, Reynolds J, Whatley M, Kurwa A, Tsokos M, Salzer W, Gillespie A, Baldwin A, Derdak J, Widemann B. 18-fluorodeoxyglucose-positron emission tomography (FDG-PET) evaluation of nodular lesions in patients with Neurofibromatosis type 1 and plexiform neurofibromas (PN) or malignant peripheral nerve sheath tumors (MPNST). Pediatr Blood Cancer. 2013 Jan;60(1):59-64. doi: 10.1002/pbc.24212. Epub 2012 May 29. PMID 22645095
- [Background] Salskov A, Tammisetti VS, Grierson J, Vesselle H. FLT: measuring tumor cell proliferation in vivo with positron emission tomography and 3'-deoxy-3'-[18F]fluorothymidine. Semin Nucl Med. 2007 Nov;37(6):429-39. doi: 10.1053/j.semnuclmed.2007.08.001. PMID 17920350
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0163.html